CLINICAL TRIAL: NCT03075215
Title: Strategic MAnagement to Optimize Response To Cardiac Resynchronization Therapy Registry (SMART Registry)
Brief Title: Strategic MAnagement to Optimize Response To Cardiac Resynchronization Therapy Registry
Acronym: SMART Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C1949
Record Dates: First submitted 2017-03-05; First posted 2017-03-09 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Device Programming of the Boston Scientific Cardiac Resynchronization Therapy Defibrillator (CRT-D) — The optimization during the standard of care visits in the first 12 months following implantation

SUMMARY:
To learn in a general Cardiac Resynchronization Therapy Defibrillators (CRT-D) population, which optimization techniques are used and how effective they are. It will compare 12-month response rates among different optimization methods and characterize which selected subject subgroups achieve better response than others.

A subset of SMART Registry subjects will contribute to the NG4 Post Market Clinical Follow Up (PMCF) Cohort whose objective is collecting data on the NG4 CRT-D features and device usage in a real world setting and monitor long term safety associated with these devices to support CE Mark.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted or upgraded with a NG3 or NG4 CRT-D device connected with any manufacturer quadripolar LV lead based on BSC labeling for devices in specific geographies.
* Subjects must be enrolled between 1 and 21 calendar days post CRT-D implantation procedure.
* Subject is age 18 or above, or of legal age to give informed consent specific to each country and national laws
* Subject is willing and capable of complying with follow-up visits and procedures as defined by this protocol

Exclusion Criteria:

* Subject with documented life expectancy of less than 12 months
* Subject currently on the active heart transplant list or has a current Left Ventricular Assist Device or other assist device (mechanical circulatory support device).
* Subject who have had a pre-existing CRT device
* Subject enrolled in any other concurrent clinical trial without prior written approval from BSC Clinical Trial Manager
* Women of childbearing potential who are or might be pregnant at time of study enrolment
* Any contra-indication to receive a CRT-D device per local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects implanted with a quadripolar NG3 or NG4 CRT-D device in conjunction with a quadripolar lead from any manufacturer will be selected based on the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2044 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Ignacio Garcia-Bolao, PhD, FESC, Principal Investigator — Clinica Universidad de Navarra
Locations (139):
- United States (29):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CardioVascular Associates of Mesa, Mesa, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Western Connecticut Health Network/ Danbury Hospital, Danbury, Connecticut
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - The University of Illinois Medical Center, Chicago, Illinois
  - Riverside Medical Center / Midwest Arrhythmia Consultants, Kankakee, Illinois
  - Ball Memorial Hospital, Muncie, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - Hurley Medical Center, Flint, Michigan
  - Summit Medical Group, P.A., Berkeley Heights, New Jersey
  - Trinity Medical WNY,PC, Buffalo, New York
  - Columbia. University Medical Center/ NY Presbyterian Hospital, New York, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Kettering Medical Center, Kettering, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Regional Cardiac Arrythmia, Washington, Pennsylvania
  - Texas Heart Rhythm, Houston, Texas
  - McAllen Medical Heart Hospital, McAllen, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
- Australia (5):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula Health, Frankston, Victoria
  - Barwon Health Myers House Ground Floor Geelong Hospital, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (3):
  - Landeskrankenhaus Salzburg Universitätsklinikum der PMU, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Univ.Klinik für Innere Medizin II, Vienna
  - Krankenhaus Nord, Vienna
- Belgium (2):
  - Virga Jesse Ziekenhuis, Hasselt
  - UCL de Mont Godinne, Yvoir
- Canada (4):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Fleurimont Hospital (CHU de Sherbrooke), Sherbrooke, Quebec
  - Royal Alexandra Hospital - Cardiology Research CK Hui Heart Centre, Edmonton
  - Hôpital du Sacré-Cœur de Montréal, Montreal
- Czechia (3):
  - Faculty Hospital U sv Anny, Brno
  - Kardiologicke centrum AGEL, Pardubice
  - IKEM - Institut klinicke a experimentalni mediciny, Prague
- France (22):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - CHU de Besancon, Besançon
  - CHU Brest - Hopital Cavale Blanche, Brest
  - Ch de Cannes, Cannes
  - APHP CHU Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - Hopital Privé de Clairval, Marseille
  - Hospital Prive Jacques Cartier, Massy
  - CH Annecy Genevois, Metz-Tessy
  - Clinique du Millénaire, Montpellier
  - NCN Nouvelles Cliniques Nantaises, Nantes
  - CHU Nimes Cedex, Nîmes
  - Chru Orleans, Orléans
  - CHG de Pau, Pau
  - CHU de Poitiers, Poitiers
  - CHU Amiens hopital sud, Salouël
  - Clinique Pasteur, Toulouse
  - CHU TOURS - Hospital Trousseau, Tours
  - Clinique Saint Gatien, Tours
  - CH Belfort Montbeliard, Trévenans
  - Hôpital Nord Franche-Comté, Trévenans
  - Centre Hospitalier de Valence, Valence
- Germany (20):
  - Charite Universitätsmedizin Berlin CBF, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Klinikum Links der Weser-Elektrophysiologie Bremen, Bremen
  - Augusta Krankenhaus, Düsseldorf
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitares Herzentrum Hamburg/Universitaetsklinik Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Oberhavel Kliniken, Hennigsdorf
  - Marien Hospital Herne, Herne
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universität Mainz zentrum fur kardiologie, Mainz
  - Klinikum Mannheim GMBH, Mannheim
  - Kliniken Maria-Hilf GmbH, Mönchengladbach
  - Deutsches Herzzentrum Muenchen, Munich
  - Krankenhaus Martha Maria, Nuremberg
  - Klinikum Oldenburg AoR, Oldenburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (15):
  - Voc Cardiologia Ospedaliera Polocino di Bari, Bari
  - Magna Graecia University AUO Mater Domini di Catanzaro, Catanzaro
  - Azienda Ospedaliero - Universitaria di Ferrara, Ferrara
  - Ospedale Vito Fazzi, Lecce
  - Federico II University of Naples, Naples
  - Ospedale Monaldi, Napoli
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedaliera di Padova, Padua
  - A.O.U. Policlinico Paolo Giaccone, Palmero
  - Ospedale Maria Paternò Arezzo, Ragusa
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale San Pietro Fatebenefratelli, Rome
  - Policlinico Casilino, Rome
  - Ospedale Santa Maria della Misericordia di Rovigo, Rovigo
  - Azienda Socio-Sanitaria Territoriale dei Sette Laghi, Varese
- Netherlands (6):
  - Noordwest Ziekenhuisgroep Alkmaar, Alkmaar
  - Amphia Ziekenhuis, Breda
  - Medisch Spectrum Twente, Enschede
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - Maasstad Hospital, Rotterdam
- Portugal (3):
  - Hospital da Senhora da Oliveira, Guimarães
  - Hospital Santa Maria (Centro Hospitalar de Lisboa Norte), Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto
- The National Institute of Cardiovascular Diseases, Bratislava, Slovakia
- Spain (13):
  - Hospital General Universitario, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Bellvitge, Barcelona
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Virgen De Las Nieves, Granada
  - Hospital Infanta Leonor, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marques De Valdecilla, Santander
  - Hospital Virgen Macarena, Seville
  - Hospital nuestra senora del prado, Talavera de la Reina
- CHUV Lausanne, Lausanne, Switzerland
- United Kingdom (12):
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - Belfast City Hospital, Belfast, Northern Ireland
  - Blackpool Teaching Hospitals NHS Foundation Trust', Blackpool
  - Bristol Heart Institute, Bristol
  - Papworth Hospital, Cambridge
  - Addenbrookes Hospital, Cambridge
  - Golden Jubilee National Hospital, Glasgow
  - LHCH (Liverpool Heart and Chest Hospital), Liverpool
  - St Bartholomews Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Northampton General Hospital, Northampton
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 2044 subjects were enrolled into the study which included 103 PMCF subjects. For 9 of those subjects (PMCF = 4) the data could not be used and 30 subjects were consent ineligible.
Groups:
- Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.: Subjects implanted de-novo with AUTOGEN, INOGEN, DYNAGEN, RESONATE HF, RESONATE, MOMENTUM, CHARISMA or VIGILANT Boston Scientific (BSC) Cardiac Resynchronization Therapy Defibrillators (CRT-D) had their CRT Response rate evaluated at 12 months, defined by the Milton Packer Clinical Composite Score (CCS). This endpoint combines four metrics: All-cause mortality, Heart failure events, NYHA Class, and Quality of life as measured with the patient global assessment instrument. A subset of 103 subjects implanted with Boston Scientific CRT-D were followed for 36 months to evaluate the PG (pulse generator) related Complication Free rate at 36 months. A SMART Registry subject was considered part of this PMCF (Post Market Clinical Follow Up) when enrolled in a European site, had an RESONATE HF, RESONATE, MOMENTUM, CHARISMA or VIGILANT BSC CRT-D implanted and Left Ventricular MultiSite Pacing (LV MSP) feature was enabled at any time during the initial 12 months follow up.
Period: 12-Month Primary Endpoint
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
Started | 2005
Completed | 1586
Not Completed | 419
Not completed — Death | 152
Not completed — Withdrawal by Subject | 267
Period: Post Market Clinical Follow-Up ONLY
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
Started | 103
Completed | 63
Not Completed | 40
Not completed — Death | 15
Not completed — Withdrawal by Subject | 25

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
Number analyzed (Participants) | 2005
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 462
  Male | 1543
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1230
  Black | 86
  Other | 17
  Race Not Disclosed | 672

OUTCOME MEASURES:

1. Primary Outcome: CRT Response Rate
Description: The traditional outcome of interest when using the Clinical Composite Score (CCS) is the proportion of patients who improved. Improvement was defined as remaining alive and free of heart failure hospitalization while also demonstrating improvement in NYHA Class, patient Global Assessment, or both. Patients were considered worsened if they died, experienced a heart failure hospitalization, or had worsened NYHA Class or patient Global Assessment. Patients who neither improved nor worsened were classified as "no change."
Time Frame: 12 months
Population: Subjects must have a complete composite score at 12 months of follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
Number analyzed (Participants) | 1558
Participants
  Improved | 918
  No Change | 312
  Worsened | 328

2. Primary Outcome: Percentage of Post Market Clinical Follow Up Participants Without NG4 Pulse Generator Related Complications
Description: Complication Free rate. PG-related Complication is defined as those detectable adverse events that resulted in:
  * Death
  * Serious injury
  * Correction of PG failure requiring invasive intervention
  * Permanent loss of PG device function. Permanent loss of device function is defined as any Pulse Generator (PG) that reverts to Safety Core or any PG rendered unable to deliver pacing or shocks Complications that are determined to be associated with the PG will be considered PGrelated complications (PG) and count against the PMCF endpoint. Complications related to the LV, RV, RA leads will not be counted against the PMCF endpoint.
Time Frame: 36 months
Population: A total of 103 subjects were classified as NG4 PMCF subjects at time of enrollment, among them 4 subjects data sets were not cleaned and unable to get corrected upon the end of the study. The final analyzed count is 99 subjects.
Measure: Number; unit: % of participants
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
Number analyzed (Participants) | 99
% of participants | 97.9

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: 2005 enrolled subjects plus 10 consent ineligible subjects with devices were considered to be at risk of AEs
Groups:
- Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.: Subjects implanted de-novo with AUTOGEN, INOGEN, DYNAGEN, RESONATE HF, RESONATE, MOMENTUM, CHARISMA or VIGILANT Boston Scientific (BSC) Cardiac Resynchronization Therapy Defibrillators (CRT-D) had their CRT Response rate evaluated at 12 months, defined by the Milton Packer Clinical Composite Score (CCS). This endpoint combines four metrics: All-cause mortality, Heart failure events, NYHA Class, and Quality of life as measured with the patient global assessment instrument. A subset of 103 subjects implanted with Boston Scientific CRT-D were followed for 36 months to evaluate the PG (pulse generator) related Complication Free rate at 36 months. A SMART Registry subject was considered part of this PMCF (Post Market Clinical Follow Up) when enrolled in a European site, had an RESONATE HF, RESONATE, MOMENTUM, CHARISMA or VIGILANT BSC CRT-D implanted and Left Ventricular MultiSite Pacing (LV MSP) feature was enabled at any time during the initial 12 months follow up. Any reportable adverse events (including deaths) from these 103 subjects, are represented in the mortality and adverse event sections of the results.
Arm/Group | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer.
All-Cause Mortality (participants affected / at risk) | 152/2015
Serious Adverse Events (participants affected / at risk) | 575/2015
Other Adverse Events (participants affected / at risk) | 132/2015
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer. (N=2015)
Hematological (Blood and lymphatic system disorders) | 9 (11)
Aortic Regurgitation (Cardiac disorders) | 2 (2)
Aortic Stenosis (Cardiac disorders) | 4 (4)
Arrhythmia-Other (Cardiac disorders) | 1 (1)
Atrial Fibrillation (AF) (Cardiac disorders) | 43 (43)
Atrial Flutter (Cardiac disorders) | 10 (10)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 13 (13)
Cardiac Medication Complication - Heart Failure (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 10 (10)
Chest Pain - Heart Failure (Cardiac disorders) | 1 (1)
Dyspnea - Heart Failure (Cardiac disorders) | 36 (40)
Gastrointestinal - Heart Failure (Cardiac disorders) | 2 (2)
Heart Failure Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 9 (9)
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 63 (74)
Hypotension - Heart Failure (Cardiac disorders) | 1 (1)
Incessant VT/ VT Storm (Cardiac disorders) | 4 (4)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 3 (3)
Multi-system Failure - Heart Failure (Cardiac disorders) | 6 (6)
Multiple Heart Failure Symptoms (Cardiac disorders) | 84 (108)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 5 (6)
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 5 (6)
Pericardial effusion - unrelated procedure/device (Cardiac disorders) | 4 (4)
Peripheral edema - Heart Failure (Cardiac disorders) | 6 (6)
Pleural Effusion - Heart Failure (Cardiac disorders) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 3 (3)
Pulmonary Edema - Heart Failure (Cardiac disorders) | 6 (6)
Pulseless Electrical Activity (PEA) (Cardiac disorders) | 1 (1)
Renal Failure/Insufficiency - Heart Failure (Cardiac disorders) | 4 (4)
Syncope - Heart Failure (Cardiac disorders) | 3 (3)
Valvular Damage/Valvular insufficiency (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (VF) (Cardiac disorders) | 9 (10)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 27 (40)
Endocrine (Endocrine disorders) | 8 (8)
Gastrointestinal (Gastrointestinal disorders) | 30 (44)
Adverse Reaction - Medication (General disorders) | 4 (4)
Chest Pain - Other (General disorders) | 7 (7)
Death (General disorders) | 34 (34)
Dizziness (General disorders) | 3 (3)
Fatigue/Weakness (General disorders) | 2 (2)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 3 (4)
Multi-System Failure (General disorders) | 5 (5)
Multiple Symptoms (General disorders) | 4 (4)
Patient Condition - Non-Cardiovascular - OTHER (General disorders) | 3 (3)
Physical Trauma (General disorders) | 17 (19)
Syncope (General disorders) | 6 (6)
Immune (Immune system disorders) | 1 (1)
Fever and/or Virus (Infections and infestations) | 1 (1)
Infection (> 30 days post implant) (Infections and infestations) | 10 (10)
Localized Infection (Infections and infestations) | 7 (8)
System Infection (Infections and infestations) | 20 (22)
Hematoma - pocket (≤ 30 days post-implant) (Injury, poisoning and procedural complications) | 4 (5)
Pneumothorax (Injury, poisoning and procedural complications) | 2 (2)
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 2 (2)
Post -Surgical infection (≤ 30 days post implant) (Injury, poisoning and procedural complications) | 2 (2)
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 1 (1)
Procedure - PG System - Other (Injury, poisoning and procedural complications) | 1 (1)
Unrelated procedure/device - OTHER (Injury, poisoning and procedural complications) | 1 (1)
Venous occlusion (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 (12)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (22)
Neurological (Nervous system disorders) | 15 (15)
Conductor Coil Fracture - RA (Product Issues) | 2 (2)
Conductor Coil Fracture - RV (Product Issues) | 1 (1)
Dislodgement - Elevated Threshold - RA (Product Issues) | 1 (1)
Dislodgement - Elevated threshold - LV (Product Issues) | 3 (4)
Dislodgement - Elevated threshold - RV (Product Issues) | 1 (1)
Dislodgement - Extracardiac stimulation - LV (Product Issues) | 3 (3)
Dislodgement - Extracardiac stimulation - RV (Product Issues) | 1 (1)
Dislodgement - Multiple signs - LV (Product Issues) | 3 (3)
Dislodgement - Multiple signs - RV (Product Issues) | 2 (3)
Dislodgement - Multiple signs- RA (Product Issues) | 2 (2)
Dislodgement - No reported signs - LV (Product Issues) | 6 (6)
Dislodgement - No reported signs - RA (Product Issues) | 4 (4)
Dislodgement - No reported signs - RV (Product Issues) | 4 (4)
Dislodgement - Unable to Capture - LV (Product Issues) | 3 (3)
Dislodgement - Unable to capture - RV (Product Issues) | 5 (5)
Electrode Damaged - RA (Product Issues) | 1 (1)
Elevated Threshold - LV (Product Issues) | 1 (1)
Elevated Threshold - RA (Product Issues) | 2 (2)
Elevated Threshold - RV 2140 - Extracardiac Stimulation - RV (Product Issues) | 5 (5)
Extracardiac Stimulation - LV (Product Issues) | 6 (7)
Helix damaged - RA (Product Issues) | 1 (1)
High Out of Range Impedance - LV (Product Issues) | 1 (1)
Impedance Out of Range (Product Issues) | 1 (1)
Inappropriate Tachy Therapy - SVT (Product Issues) | 2 (2)
Inappropriate tachy therapy - SVT (Product Issues) | 3 (3)
Inappropriate tachy therapy - Other (Product Issues) | 1 (1)
Other Lead Related (Product Issues) | 1 (1)
PG System diagnosis - OTHER (Product Issues) | 1 (1)
PG System - Patient Related - OTHER (Product Issues) | 3 (3)
Unable to Capture - LV (Product Issues) | 1 (1)
Unable to Capture - RV (Product Issues) | 2 (2)
Unable to Capture - RA (Product Issues) | 1 (1)
Psychological (Psychiatric disorders) | 2 (2)
Genitourinary (Renal and urinary disorders) | 10 (12)
Renal (Renal and urinary disorders) | 30 (36)
Adverse Reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural Effusion - unrelated procedure/device (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax - unrelated procedure/device (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 35 (47)
Integumentary (Skin and subcutaneous tissue disorders) | 4 (4)
Skin burns (Skin and subcutaneous tissue disorders) | 1 (1)
Cerebrovascular Accident (CVA) (Vascular disorders) | 3 (3)
Cerebrovascular accident (CVA) - ischemic (Vascular disorders) | 6 (6)
Chest Pain - Ischemic (Vascular disorders) | 6 (6)
Coronary Artery Disease (Vascular disorders) | 16 (17)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 3 (3)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 4 (4)
Myocardial Infarction (Vascular disorders) | 9 (10)
Peripheral Vascular Disease (Vascular disorders) | 11 (12)
Pulmonary Embolism (PE) (Vascular disorders) | 5 (5)
Transient Ischemic Attack (TIA) (Vascular disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted De-novo With a BSC CRT-D Together With a Quadripolar Lead From Any Manufacturer. (N=2015)
Atrial (Type I) Flutter (Cardiac disorders) | 2 (2)
Atrial Fibrillation (AF) (Cardiac disorders) | 16 (18)
Atrial Flutter (Cardiac disorders) | 3 (3)
Atrial Tachycardia/Other SVT (e.g. AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3)
Dyspnea - Heart Failure (Cardiac disorders) | 13 (16)
Heart Failure Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 2 (3)
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 6 (9)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 1 (1)
Multiple Heart Failure Symptoms (Cardiac disorders) | 7 (8)
Patient Condition - Cardiovascular - OTHER (Cardiac disorders) | 1 (1)
Pericardial Effusion - Heart Failure (Cardiac disorders) | 1 (1)
Peripheral edema - Heart Failure (Cardiac disorders) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 2 (2)
Torsades de Pointes (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (VF) (Cardiac disorders) | 5 (7)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 17 (17)
Chest Pain - Other (General disorders) | 3 (3)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Syncope (General disorders) | 2 (2)
Vasovagal Reaction (General disorders) | 1 (1)
Infection (> 30 days post implant) (Infections and infestations) | 1 (1)
System Infection (Infections and infestations) | 1 (1)
Post Surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 1 (1)
Post-surgical pocket hemorrhage/bleeding/drainage (Injury, poisoning and procedural complications) | 1 (1)
Thromboembolic events (Injury, poisoning and procedural complications) | 1 (1)
Venous occlusion (Injury, poisoning and procedural complications) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Conductor Coil Fracture - RA (Product Issues) | 1 (1)
Dislodgement - Elevated threshold - RV (Product Issues) | 1 (1)
Dislodgement - Multiple signs - LV (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Dislodgement - No reported signs - LV (Product Issues) | 1 (1)
Elevated Threshold - LV (Product Issues) | 1 (1)
Elevated Threshold - RA (Product Issues) | 1 (1)
Elevated Threshold - RV 2140 - Extracardiac Stimulation - RV (Product Issues) | 2 (2)
Extracardiac Stimulation - LV (Product Issues) | 20 (21)
Inappropriate Tachy Therapy - SVT (Product Issues) | 1 (1)
Inappropriate tachy therapy - SVT (Product Issues) | 4 (4)
Inappropriate tachy therapy - NSR (Product Issues) | 2 (2)
Inappropriate tachy therapy - Other (Product Issues) | 1 (1)
Other - PG System (Product Issues) | 1 (1)
Oversensing - RA (Product Issues) | 1 (1)
Pacemaker Mediated Tachycardia (PMT) (Product Issues) | 5 (5)
Renal (Renal and urinary disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations include a lack of a control group, but a non-randomized observational study with 2005 subjects is appropriate to meet the study's objectives to obtain "real world" therapy outcome. Due to COVID-19, there was an increase in missed visits/withdrawals, the impact to the data was minimal, 75.8% of 12-month visits were before March 2020 and there was sufficient data to power the 36-month analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Sponsor may extend the review period for another 90 days to take steps to protect its intellectual property interests, or to remove any language detrimental to Sponsor's intellectual property interests.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03075215/Prot_SAP_000.pdf